CLINICAL TRIAL: NCT01821352
Title: A Double-Blind, Placebo-Controlled Randomized Evaluation of the Effect of the Erchonia Obesity Laser on the Reduction of Circumference of the Hips, Waist and Upper Abdomen for Individuals With a Body Mass Index (BMI) of 30 to 40 kg/m2
Brief Title: Study of Low Level Laser Therapy to Reduce Body Circumference in Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC_OL_001
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erchonia Obesity Laser (Active Comparator): The Erchonia® Obesity Laser is made up of 10 independent 17 milliWatts (mW), 532 nanometer (nm) green laser diodes, each diode positioned 120 degrees apart from the next with each titled at a 30 degree angle. The Erchonia® Obesity Laser is a pulsed wave variable frequency device.
  Interventions: Device: Erchonia Obesity Laser
- Placebo Laser (Placebo Comparator): Laser device emitting sham green light that has no therapeutic effect.
  Interventions: Device: Placebo Laser

INTERVENTIONS:
Device: Erchonia Obesity Laser — 10 independent 17 milliwatts 532 nm green diode lasers
  Arms: Erchonia Obesity Laser
Device: Placebo Laser — Emits light that has no therapeutic effect
  Arms: Placebo Laser

SUMMARY:
The purpose of this study is to determine whether low level laser light therapy is effective in reducing circumference of the waist, hips and upper abdomen in obese individuals.

DETAILED DESCRIPTION:
The American Society of Plastic Surgeons (ASPS) 2011 report states that the market for cosmetic procedures has shown significant growth over the past two years, with 13.8 million cosmetic plastic surgery procedures performed in the United States in 2011, up 5% since 2010. While surgical cosmetic procedures did increase significantly from 2010 to 2011, the overall growth in cosmetic procedures is being primarily driven by a substantial rise in minimally-invasive procedures. Cosmetic minimally-invasive procedures increased 6%, with nearly 12.2 million cosmetic minimally-invasive procedures having been performed in 2011. This highlights the growing consumer demand for non- or minimally-invasive cosmetic procedures that do not involve surgical procedures such as liposuction and the associated risks, potential complications and lengthy and painful recovery processes.

Low level laser light therapy, such as that to be provided through application of the Erchonia® Obesity Laser in this clinical study protocol, offers a simple, non-invasive, safe, effective and side-effect free alternative to achieving body circumference reduction.

Justification for this assertion of anticipated safety and effectiveness of the application of the Erchonia® Obesity Laser for the reduction of body circumference is found through three FDA clearances for Erchonia® Low Level Laser devices for body circumference reduction indications, as follows:

K123237 (532 nm green light diodes): Erchonia® Zerona™ 2.0 Laser: is indicated for use as a non-invasive dermatological aesthetic treatment as an adjunct for individuals intending to undergo liposuction procedures for the reduction of circumference of hips, waist, and thighs.

K121695 & K082609 (635 nm red light diodes): Erchonia® ML Scanner (MLS) & Erchonia® Zerona: is indicated for use as a non-invasive dermatological aesthetic treatment as an adjunct for individuals intending to undergo liposuction procedures for the reduction of circumference of hips, waist, and thighs.

K121690 & K120257 (635 nm red light diodes): Erchonia® MLS, Zerona, Zerona-AD: is indicated for use as a non-invasive dermatological aesthetic treatment as an adjunct for individuals intending to undergo liposuction procedures for the reduction of circumference of the upper arms.

Therefore, Erchonia low level lasers have been determined safe and effective by the FDA for application for body circumference reduction indications for multiple body areas, such that evaluation of application of the Erchonia Obesity Laser to reducing body circumference in more overweight individuals is a natural extension of its proven and accepted application for body circumference reduction purposes.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) is between 30 kg/m² and 40 kg/m², inclusive.
* Subject indicated for liposuction or use of liposuction techniques for the removal of localized deposits of adipose tissues that do not respond to diet and exercise; specifically for the indication of body contouring in the areas of the hips, waist and upper abdomen. (As per the American Academy of Cosmetic Surgery's 2006 Guidelines for Liposuction Surgery developed by A joint Ad Hoc Committee of the American Society of Lipo-Suction Surgery (ASLSS) and the American Academy of Cosmetic Surgery (AACS))
* Subject is willing and able to abstain from partaking in any treatment other than the study procedure (existing or new) to promote body contouring/ circumference reduction/weight loss during the course of study participation.
* Subject is willing and able to maintain his or her regular (typical pre-study) diet and exercise regimen without effecting significant change in either direction during study participation

Exclusion Criteria:

* Body Mass Index (BMI) is less than 30 kg/m² or greater than 40 kg/m².
* Known cardiovascular disease such as cardiac arrhythmias, congestive heart failure.
* Cardiac surgeries such as cardiac bypass, heart transplant surgery, pacemakers.
* Prior surgical intervention for body sculpting/weight loss, such as liposuction, abdominoplasty, stomach stapling, lap band surgery, etc.
* Medical, physical, or other contraindications for body sculpting/weight loss.
* Current use of medication(s) known to affect weight levels/cause bloating or swelling and for which abstinence during the course of study participation is not safe or medically prudent.
* Any medical condition known to affect weight levels and/or to cause bloating or swelling.
* Diagnosis of, and/or taking medication for, irritable bowel syndrome.
* Active infection, wound or other external trauma to the areas to be treated with the laser.
* Known photosensitivity disorder.
* Current active cancer or currently receiving treatment for cancer.
* Pregnant or planning pregnancy prior to the end of study participation.
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in past two years.
* Developmental disability or cognitive impairment that in the opinion of the investigator would preclude adequate comprehension of the informed consent form and/or ability to record the necessary study measurements.
* Involvement in litigation and/or a worker's compensation claim and/or receiving disability benefits related to weight-related and/or body shape issues.
* Participation in a clinical study or other type of research in the past 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Shanks, Study Director — Erchonia Corporation
Locations (2):
- United States (2):
  - Surgeons Inc., Noblesville, Indiana
  - Bloomfield Laser and Cosmetic Surgery Center, Bloomfield Hills, Michigan

REFERENCES:
- [Derived] Roche GC, Shanks S, Jackson RF, Holsey LJ. Low-Level Laser Therapy for Reducing the Hip, Waist, and Upper Abdomen Circumference of Individuals with Obesity. Photomed Laser Surg. 2017 Mar;35(3):142-149. doi: 10.1089/pho.2016.4172. Epub 2016 Dec 9. PMID 27935737

RESULTS

PARTICIPANT FLOW:
Groups:
- Erchonia Obesity Laser: The Erchonia® Obesity Laser is made up of 10 independent 17 milliWatts (mW) 532 nanometer (nm) green laser diodes, each diode positioned 120 degrees apart from the next with each titled at a 30 degree angle. The Erchonia® Obesity Laser is a pulsed wave variable frequency device.
- Placebo Laser: Placebo Laser device emits sham green light that has no therapeutic effect.
Period: Overall Study
Arm/Group | Erchonia Obesity Laser | Placebo Laser
Started | 28 | 25
Completed | 28 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Laser: Placebo Laser device emitting sham green light that has no therapeutic effect.
- Total: Total of all reporting groups
Arm/Group | Erchonia Obesity Laser | Placebo Laser | Total
Number analyzed (Participants) | 28 | 25 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.32 (10.91) | 47.84 (9.30) | 47.04 (10.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 45
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 23 | 19 | 42
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 25 | 53
Total Circumference Measurement [Mean (Standard Deviation); unit: inches] — Circumference of the hips, waist and the upper abdomen was measured in inches (in) at standardized locations using a flexible tape measure. The 3 individual area circumference measurements were added to attain a total body circumference measurement in inches.
  inches | 123.35 (10.29) | 122.81 (11.85) | 123.04 (10.95)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Body Mass Index (BMI) was calculated as kilograms per meter squared (kg/m2).
  kg/m2 | 34.58 (3.06) | 33.60 (2.98) | 34.04 (3.02)

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Proportion of Primary Outcome Successes Between Treatment Groups for Change in Combined Circumference Measurements
Description: Individual measurements in inches of the waist, hips and upper abdomen were combined to calculate a total body circumference measurement. Change in combined circumference measurement from baseline to 4 weeks was calculated for each subject. Individual subject success was defined as a change of 3.0 inches or more in the combined circumference measurement across the evaluation period. A decrease in combined circumference measurement is positive for individual subject success. An increase in combined circumference measurement is negative for individual subject success. Overall study success was defined as a 40% or greater difference between the proportion of individual successes in each treatment group.
Time Frame: Baseline and 4 Weeks
Measure: Number; unit: participants
Arm/Group | Erchonia Obesity Laser | Placebo Laser
Number analyzed (Participants) | 28 | 25
participants | 20 | 3
Statistical Analysis 1: Comparison: Erchonia Obesity Laser vs Placebo Laser; Test type: Superiority or Other; p < 0.00005, Fisher Exact

2. Other Pre Specified Outcome: Subject Satisfaction With Procedure Outcome
Description: Subjects rated satisfaction with the outcome of the study procedures with respect to change in body shape on the following 5-point scale: Very Satisfied, Somewhat Satisfied, Neither Satisfied nor Dissatisfied, Not Very Satisfied, Not at All Satisfied.
  Results are reported as the number of subjects in each treatment group who rated study outcome satisfaction as 'Very Satisfied' or 'Somewhat Satisfied'.
Time Frame: 4 Weeks
Measure: Number; unit: participants
Arm/Group | Erchonia Obesity Laser | Placebo Laser
Number analyzed (Participants) | 28 | 25
participants | 22 | 4
Statistical Analysis 1: Comparison: Erchonia Obesity Laser vs Placebo Laser; Test type: Superiority or Other; p < 0.0001, Fisher Exact

3. Primary Outcome: Change in Combined Circumference Measurement
Description: Individual measurements in inches of the waist, hips and upper abdomen were combined to calculate a total combined body circumference measurement. Change in combined circumference measurement is calculated as the difference in circumference measurements from baseline to endpoint (4 weeks). A negative (-) change indicates a decrease in circumference and is positive for study success. A positive (+) change indicates an increase in circumference and is negative for study success.
Time Frame: Baseline and 4 Weeks
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Erchonia Obesity Laser | Placebo Laser
Number analyzed (Participants) | 28 | 25
inches | -4.14 (2.99) | -0.71 (1.26)
Statistical Analysis 1: Comparison: Erchonia Obesity Laser vs Placebo Laser; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 Weeks
Arm/Group | Erchonia Obesity Laser | Placebo Laser
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/25
Other Adverse Events (participants affected / at risk) | 0/28 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No